CLINICAL TRIAL: NCT07071727
Title: Short Course Of Preoperative Radiotherapy in Head and Neck-, Trunk- and Extremity Soft Tissue Sarcomas; a Second Randomized Phase II Clinical Trial
Brief Title: Short Course of Radiotherapy Prior to Surgery of Soft Tissue Sarcomas
Acronym: SCOPES II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Institute of Oncology in Warsaw (Unknown); Radboud University Medical Center (Other); University Medical Center Groningen (Other); Leiden University Medical Center (Other); Amsterdam UMC (Other); Erasmus Medical Center (Other); Maastro (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M24SCT; NL009842 (Other: Centrale Commissie Mensgebonden Onderzoek)
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Sarcoma of Soft Tissue; Sarcoma; Sarcoma, Soft Tissue
Keywords: preoperative radiotherapy; radiotherapy
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Intervention Model Description: Randomization between two study arms: arm A of 14 x 3 Gy in 3 weeks and arm B of 5 x 6 Gy in one week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Other): Arm A: Preoperative radiotherapy to a total dose of 42 Gy in 14 once daily fractions of 3 Gy, in an overall treatment time of three weeks.
  Interventions: Radiation: Preoperative radiotherapy
- Arm B (Other): Arm B: Preoperative radiotherapy to a total dose of 30 Gy in 5 once daily fractions of 6 Gy, in an overall treatment time of one week.
  Interventions: Radiation: Preoperative radiotherapy

INTERVENTIONS:
Radiation: Preoperative radiotherapy — preoperative radiotherapy

SUMMARY:
Based upon the preliminary data derived from first SCOPES clinical trial and the results of patients treated during the recent COVID-19 pandemic, patients with soft tissue sarcomas (STS) can be preoperatively irradiated in a modestly hypofractionated schedule of 14 x 3 Gy. From a toxicity and efficacy point of view, this regimen equals the outcomes after a conventionally fractionated regimen of 25 x 2 Gy in five weeks. Moreover, the rationale for investigating (modest) hypofractionation in the clinic comes both from a logistic point of view (patient convenience and a lower pressure on radiotherapy equipment), form prior phase II clinical evidence and from (cellular) radiobiological observations. There is phase II trial evidence suggesting that even more (ultra-) hypofractionation to 5 x 6 Gy is also safe and effective. Within this study, patients will be randomized to receive either the modestly hypofractionated conventional schedule of 14 x 3 Gy or an even shorter preoperative regimen of 5 x 6 Gy, in the hypothesis that both the postoperative wound complication rate until 120 days after surgery, as well as the local control probability at two years are comparable in both arms.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed intermediate to high grade soft tissue sarcoma localized to the head and neck area, to the trunk and chest wall or to the extremities, for which the standard treatment is a combination of and radiotherapy and surgery (deep seated and/or ≥ 5cm in largest tumor diameter and/or an anticipated close resection margin and/or grade II/III according to the FNCLCC definition);
* Absence of regional and/or distant disease. Patients must be staged by at least a CT scan of the chest. Staging may also be performed by FDG-PET scanning and/or total body MRI scans;
* WHO Performance Status ≤ 2;
* Able and willing to undergo preoperative radiotherapy;
* Able and willing to undergo definitive surgery;
* Able and willing to comply with regular follow-up visits;
* Able and willing to complete patient reported outcome questionnaires (health-related quality of life and cost effectiveness);
* Able and willing to undergo randomization;
* Age ≥ 18 years;
* Signed written informed consent.

Exclusion Criteria:

* Prior malignancies; except another malignancy and disease-free for ≥ 5 years, or completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma;
* Patients with locally recurrent sarcomas, regardless of the management of the first sarcoma diagnosis;
* Ewing sarcoma and other PNET family tumors, rhabdomyosarcomas (both pediatric and adult), osteosarcomas;
* Myxoid liposarcomas, because they have shown to be exquisitely sensitive to a lower dose of radiation as compared to the 2 regimens tested in this trial.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial;
* Female patients who are pregnant;
* Intention to perform an isolated limb perfusion, instead of a tumor resection;
* Neoadjuvant chemotherapy both before and after radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2033-11-01 (Estimated)

PRIMARY OUTCOMES:
The short-term toxicity | within 120 days post-surgery
  wound complications

SECONDARY OUTCOMES:
Local control | During follow up (5 years)
  local failure after surgery
Long-term toxicity | During follow-up (5 years)
  fibrosis, edema, joint stiffness and bone fractures
Not operated patients | During follow-up (5 years)
  Outcome of patients that were irradiated per randomization but eventually were not operated upon in conjunction to the reasons why the operation was not executed

CONTACTS AND LOCATIONS:
Locations (6):
- Netherlands (6):
  - Netherlands Cancer Institute, Amsterdam
  - AUMC, Amsterdam
  - UMCG, Groningen
  - LUMC, Leiden
  - Maastro, Maastricht
  - RadboudUMC, Nijmegen

IPD SHARING:
Plan to Share IPD: Undecided